CLINICAL TRIAL: NCT06685172
Title: Comparison of the Acute Effects of Focused and Radial ESWT on Pain and Balance Performance in Individuals With Plantar Fasciitis: A Randomized Clinical Trial
Acronym: ESWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tuğba Kocahan, Associate Professor MD, Gulhane Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/285; Health Sciences University (Other: Gülhane Training and Research Hospital)
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Plantar Fascitis; Pain
Keywords: Balance; pain; plantar fasciitis; stability
MeSH Terms: conditions — Pain; Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: A total of 40 patients with plantar fasciitis were randomly assigned to focal-ESWT treatment (n= 20) or radial-ESWT treatment (n= 20).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- f-ESWT Group (Active Comparator): Twenty patients with plantar fasciitis received f-ESWT treatment once a week for four weeks.
  Interventions: Other: f-ESWT
- r-ESWT Group (Active Comparator): Twenty patients with plantar fasciitis received r-ESWT treatment once a week for four weeks.
  Interventions: Other: r-ESWT

INTERVENTIONS:
Other: f-ESWT — In the f-ESWT group, a total of 8 Hz, 0.28 mJ/mm2, and 2000 pulses were applied while in the r-ESWT group, a total of 8 Hz, 1.8 bar, and 2000 pulses were applied
  Arms: f-ESWT Group
Other: r-ESWT — In the f-ESWT group, a total of 8 Hz, 0.28 mJ/mm2, and 2000 pulses were applied while in the r-ESWT group, a total of 8 Hz, 1.8 bar, and 2000 pulses were applied
  Arms: r-ESWT Group

SUMMARY:
This study aimed to compare the acute effects of focused and radial ESWT on pain and balance performance in individuals with plantar fasciitis.

DETAILED DESCRIPTION:
This study aimed to compare the acute effects of focused and radial ESWT on pain and balance performance in individuals with plantar fasciitis. The study included 40 individuals (27 females and 13 males) aged between 18 and 63 years, presenting with plantar fasciitis (PF). Extracorporeal shockwave therapy (ESWT) was administered once a week for four weeks. The participants were randomly assigned to two groups (f-ESWT and r-ESWT). Pain levels were assessed using the Visual Analogue Scale, while Static and Dynamic Balance were evaluated using the Biodex Balance System.

ELIGIBILITY:
Inclusion Criteria:

unilateral or bilateral tenderness in the medial tubercle of calcaneus and heel pain in the first few steps in the morning, which gets worse with increased activity, absence of any known systemic disease, absence of any surgical procedure to lower extremity, absence of any treatment for PF in the last 6 months, 18-65 years, and consent to participate in the study.

Exclusion Criteria:

pregnancy, pacemaker, receiving anticoagulant therapy, uncontrolled cardiovascular disease, tumor, acute infection, nerve root compression, local dermatological or neurological problems, diabetes mellitus, taking anti-inflammatory drugs during treatment, or incomplete follow-up.

Ages: 18 Months to 63 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) was used to determine the intensity of pain in patients with PF, and Biodex Balance System device (Biodex Balance System SD, 2009 USA) was used to assess balance performance. | Baseline and 5 weeks
  The Visual Analogue Scale (VAS) was employed to ascertain the intensity of pain experienced by the affected/more affected extremities. The Biodex Balance System device (Biodex Balance System SD, 2009 USA) was used to assess balance performance.

CONTACTS AND LOCATIONS:
Overall Officials: Aydan Örsçelik, Associate Professor MD, Study Chair — Health Sciences University, Gulhane Training and Research Hospital
Locations (1):
- University of Health Sciences, Gulhane Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared after publication as an article
Supporting Information: SAP
Time Frame: Once published as an article, data can be shared for one year
Access Criteria: After the article is published, it can be requested from the responsible researcher upon request.